CLINICAL TRIAL: NCT06710639
Title: Effects of a Cognitive Training Program on Chemotherapy-induced Cognitive Impairment (Chemobrain) in Oncology Patients With Colon Cancer Undergoing Active Treatment: A Randomized Controlled Trial
Brief Title: Effects of Cognitive Training on Chemotherapy-Induced Cognitive Impairment in Colon Cancer Patients Undergoing Treatment(Chemobrain) in Oncology Patients With Colon Cancer Undergoing Active Treatment
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, Prof. Dr. Eduardo J Fernández Rodríguez, Professor, University of Salamanca
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHEMOBRAIN COLON
Record Dates: First submitted 2024-11-13; First posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Oncology; Cancer-related Cognitive Impairment; Cognitive Training; Everyday Cognition; Clinical Trials; Colon Cancer
Keywords: Oncology; Cancer-related cognitive impairment; Cognitive training; Everyday cognition; Clinical trials; Colon cancer
MeSH Terms: conditions — Neoplasms; Colonic Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health Education Program (Active Comparator): Instructions and recommendations will be provided in an informational leaflet to encourage an active and healthy lifestyle, promoting self-care and good health practices. This leaflet will include the new WHO guidelines recommending specific measures to reduce the risk of cognitive impairment. These measures are: eating healthy foods, engaging in physical activity, maintaining social contact, doing challenging cognitive games, getting good sleep, managing stress, staying hydrated, and avoiding smoking and excessive alcohol consumption.
  Interventions: Behavioral: Health Education Program
- Cognitive Training Program (Experimental): The cognitive training program (CT) focused on everyday cognition (EC) will be conducted individually. Each participant will receive a dossier specifically designed for the study. The intervention will consist of four training periods over 4 months (Period 1, P1; Period 2, P2; Period 3, P3; Period 4, P4), with 20 activities in each period. Each period will last one month (with 5 activities per week). To ensure compliance and therapeutic adherence, two types of follow-up will be carried out: in-person or via telematic (video call).
  Interventions: Behavioral: Cognitive Training Program

INTERVENTIONS:
Behavioral: Health Education Program — Instructions and recommendations will be provided in an informational leaflet to encourage an active and healthy lifestyle, promoting self-care and good health practices. This leaflet will include the new WHO guidelines recommending specific measures to reduce the risk of cognitive impairment.
  Arms: Health Education Program
Behavioral: Cognitive Training Program — The cognitive training program (CT) focused on everyday cognition (EC) will be conducted individually. Each participant will receive a dossier specifically designed for the study.
  Arms: Cognitive Training Program

SUMMARY:
Introduction: With the increasing survival rate in colon cancer, as a result of technological and biomedical advancements, it is essential to thoroughly study the secondary symptoms related to the oncological disease process. One of the most common and underestimated symptoms is cancer-related cognitive impairment (CRCI).

Objective: To evaluate the efficacy of a cognitive training program in controlling CRCI in individuals with colon cancer undergoing active treatment.

Methodology: A randomized controlled clinical trial with two parallel groups: an intervention group (IG) and a control group (CG). The study population will include individuals newly diagnosed with colon cancer. A sample size of 50 participants has been estimated, with 25 in each group, to detect a difference of 2.95 points or more in the MoCA cognitive impairment questionnaire. All participants will receive an educational leaflet based on the new WHO guidelines, which recommend specific measures to reduce the risk of cognitive impairment. In addition to receiving this informational leaflet, the IG will participate in a cognitive training program (CT) focused on everyday cognition (EC) individually. Each participant will receive a dossier with 80 intervention sessions divided into four training periods (P1-P4), each containing 20 activities. Each period will last for one month. Baseline and 4-month post-intervention evaluations will be conducted for both groups, measuring sociodemographic and clinical variables, as well as study-related cognitive impairment variables: Cognitive function (MoCA test), Everyday Cognition (PECC), Anxiety (Hamilton), Functionality (LB), Sleep Quality (PSQI), Quality of Life (ECOG), and Subjective Memory Complaints (FACT-COG).

Impact: The results of this study could lead to the design of specific cognitive interventions and the establishment of protocols for colon cancer patients undergoing active treatment, helping them manage one of the most underestimated symptoms in this patient population-CRCI-whose incidence is increasing due to the improved survival rates in this disease.

ELIGIBILITY:
Inclusion Criteria:

Being an adult (18 years or older). Having a recent pathological diagnosis of newly diagnosed colon cancer and starting oncological treatment.

Being fully capable of performing daily functions. Willingness to voluntarily participate in the study and signing the informed consent.

Exclusion Criteria:

Lack of literacy skills or significant language comprehension deficits. Having a diagnosis of a Central Nervous System tumor or participating in another cognitive stimulation program.

Having a clinical diagnosis of a neurocognitive disorder as defined in the DSM-V.

Withdrawal Criteria:

Dropping out of the program or not completing the final evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Cognitive Function | Baseline; "4 months final";
  The Montreal Cognitive Assessment Test (MoCA test) Version 8.3" (17): This test allows the detection of mild cognitive impairment (MCI) by evaluating executive functions, attention, abstraction, memory, calculation, and orientation. The administration time is 10 minutes. The maximum score is 30 points, with scores below 26 indicating MCI.
Subjective Perception of Cognitive Impairment in Oncology Patients | Baseline; "4 months final";
  FACT-COG (Version 3)" (24): This 37-item questionnaire is divided into six cognitive domains: memory, concentration, mental acuity, verbal fluency, functional interference, and multitasking ability. Additionally, the tool includes two other subscales: "notability" (comments from others) and "impact of perceived cognitive impairment on quality of life." Respondents indicate the frequency of each occurrence during the 7 days prior to the test on a 5-point Likert scale ranging from 0, "never," to 4, "several times a day." The individual subscale scores are summed to determine the total FACT-Cog score, which ranges from 0 to 148, with higher scores indicating better cognitive functioning.

SECONDARY OUTCOMES:
Everyday Cognition | Baseline; "4 months final";
  Test for the Evaluation of Everyday Cognition (PECC)" (18): This test measures individuals' ability to solve 12 real-life situations grouped into the following areas: medication management, administrative management, financial management, meal preparation, transportation, and shopping. It helps assess functional capacity in daily life. The administration time is 35 minutes.
Anxiety | Baseline; "4 months final";
  Hamilton Anxiety Rating Scale" (19): A clinical assessment tool used to evaluate the level of anxiety experienced by a person. It consists of 14 items, each with five response options ranging from "not present" to "very severe," with a score assigned to each response. A total score of 17 or less indicates mild anxiety; 18 to 24 indicates moderate anxiety; and 25 to 30 indicates severe anxiety.
Functionality | Baseline; "4 months final";
  Lawton and Brody Instrumental Activities of Daily Living Scale" (20): Designed to assess autonomy in instrumental activities in the elderly population. The administration time is 4 minutes, and each item is scored as 0 or 1, with a total score of 8.
Sleep Quality | Baseline; "4 months final";
  Pittsburgh Sleep Quality Index (PSQI)" (21): Developed to measure sleep quality in individuals aged 24 to 83 years. The administration time is 5-10 minutes. Nineteen individual items generate seven "component" scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction.
Subjective Memory Failures | Baseline; "4 months final";
  Everyday Memory Failures Questionnaire" (23): This questionnaire includes categories of forgetfulness such as "speaking, reading, and writing," "names and faces," "actions," and "learning new things." Responses are given on a Likert scale with nine response options for each question, ranging from "Never in the past 3 months" to "More than once a day." However, due to the difficulty of the nine options, other authors have used fewer response choices.

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon request in the GREDOS scientific repository of the University of Salamanca once the study is completed. Link: https://gredos.usal.es/handle/10366/3823.
Supporting Information: Study Protocol, ICF, CSR
Access Criteria: The data will be available upon request in the GREDOS scientific repository of the University of Salamanca once the study is completed. Link: https://gredos.usal.es/handle/10366/3823.
URL: http://gredos.usal.es/

DOCUMENTS (1):
  • Informed Consent Form (2024-09-01): https://cdn.clinicaltrials.gov/large-docs/39/NCT06710639/ICF_000.pdf